CLINICAL TRIAL: NCT02434991
Title: Sensorimotor Dysfunction in Achalasia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karthik Ravi, M.D., Karthik Ravi, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-009073
Record Dates: First submitted 2015-04-06; First posted 2015-05-06 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Achalasia
Keywords: trouble swallowing; food sticking; Achalasia
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Barostat (Experimental): The barostat (a thin tube, with a deflated balloon attached at the end) will be placed through your mouth down your esophagus (swallowing tube) to where your stomach and esophagus meet. The 10-cm long balloon will then be inflated with step by step pressure increases of 4mmHg for 30 seconds each to a maximum pressure of 50mmHg. The patient will rate discomfort during each step of inflation
  Interventions: Device: Barostat

INTERVENTIONS:
Device: Barostat — * During this study, the investigators will ask you to fill out questionnaires about your swallowing, chest pain, and heartburn. The investigators hope the patient will answer all of the questions, but patients can skip any questions they do not want to answer. The questionnaires will take about 15 minutes to complete.
  * A urine pregnancy test for females of childbearing years.
  * Patients will be asked to fast overnight (nothing to eat or drink for 8 hours) prior to the barostat test.
  * At this point healthy controls have completed the study.
  * Patients with achalasia will then undergo treatment for achalasia at the discretion of the primary clinician managing their case.
  * Patients will be contacted to complete a phone survey 3 & 6 months and 2 & 4 years after treatment.
  Other Names: Sensorimotor dysfunction

SUMMARY:
This study is being done to assess the esophageal muscle (swallowing tube) in patients with and without achalasia to further understand and help direct the treatment for patients with achalasia.

DETAILED DESCRIPTION:
Achalasia is currently defined solely on the basis of esophageal manometry. However, this fails to assess sensory function which may relate more to symptoms such as chest pain and heartburn. To date, the importance of sensory dysfunction in achalasia is poorly understood. The investigators want to define the relationship between esophageal sensory and motor dysfunction and symptoms in achalasia.

Following standard diagnostic evaluation including esophagogastroduodenoscopy (EGD), barium esophagram, and esophageal manometry, symptoms will be assessed utilizing a standardized questionnaire. The subjects will then undergo transoral placement of an esophageal barostat. Following a standard protocol of esophageal distension, esophageal body compliance will be recorded with esophageal body pressure and volume. Mechanosensitivity will then be assessed utilizing a stepwise esophageal distension, with patients reporting symptoms utilizing a Likert scale. Patients will then undergo conventional achalasia treatment with either pneumatic dilation or Heller myotomy at the discretion of the treating gastroenterologist. Thereafter patients will be followed via a standardized phone survey at 3 months, 6 months, 2 years, and 4 years after treatment to assess symptoms and treatment response. Patients will have standard clinical follow ups, including barium esophagram, at 1 year, 3 years, and 5 years following treatment. Outcomes: From 100 new patients with achalasia seen yearly at Mayo, the investigators anticipate recruitment of 40 eligible patients over 12 months and 10 healthy volunteers. The correlation between mechanosensitivity and esophageal body compliance with symptoms such as dysphagia, chest pain, and heartburn will be measured in Types I, II and III achalasia. The association of these parameters with conventional manometrically defined achalasia subtypes will also be measured. Finally, the relationship between sensorimotor dysfunction in achalasia and therapeutic outcomes will be assessed with development of predictive models to assess symptomatic outcome by barostat measurements.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-90
* Patients with achalasia, defined by an esophageal manometry study consistent with the diagnosis

Exclusion Criteria:

* Patients with EGD or esophagram findings suggestive of pseudoachalasia
* Previous history of pneumatic dilation, Heller myotomy, or botulinum toxin injection to the distal esophagus
* Esophageal diameter greater than 6 cm
* Previous history of upper gastrointestinal surgery
* Medical conditions such as severe heart or lung disease that preclude safe performance barostat
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Presence of discomfort during barostat | 20 minutes
  During each distention, patients would report presence of discomfort as: 0) none 1) sensation without discomfort 2) mild discomfort 3) moderate discomfort 4) pain. This scale has been utilized in previous studies assessing esophageal mechanosensitivity.

SECONDARY OUTCOMES:
symptoms (followup phone survey) | 3, 6 months, 2, 4 years
  Measuring symptoms (dysphagia, regurgitation, chest pain, nocturnal cough) with modified Eckardt Score 0 None 1 occasional 2 daily
  None Occasional Daily

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ravi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States